CLINICAL TRIAL: NCT02031432
Title: An Open-label, Multi-site Trial to Describe the Safety and Tolerability of Oral Cebranopadol Administered for 26 Weeks in Subjects With Cancer-related Pain Who Have Completed Treatment in the KF6005/07 Trial
Brief Title: CORAL XT - Open-label Extension Trial of the CORAL Trial
Acronym: CORAL XT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF6005/09; 2013-001877-26 (EudraCT Number); U1111-1144-0778 (Other: World Health Organization)
Record Dates: First submitted 2013-12-12; First posted 2014-01-09 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pain; Neoplasms; Chronic Pain
Keywords: cancer-related pain; cebranopadol
MeSH Terms: conditions — Pain; Neoplasms; Chronic Pain; Cancer Pain | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cebranopadol (Experimental): Cebranopadol 200 µg to 1000 µg per taken taken once a day in the morning.
  Allowed dose levels in the Maintenance Phase were 200, 400, 600, 800, or 1000 µg per day.
  Interventions: Drug: Cebranopadol

INTERVENTIONS:
Drug: Cebranopadol — Film-coated tablet; strengths: 200, 400, or 600 µg
  Other Names: GRT6005

SUMMARY:
The purpose of this trial was to find out how well cebranopadol is tolerated and how often, and which, adverse reactions occur when it is taken every day for a longer period of time. In addition, information was collected how cebranopadol affects pain and well-being in patients suffering from cancer-related pain.

DETAILED DESCRIPTION:
The trial consisted of 3 phases: Titration Phase, Maintenance Phase, and Follow-Up. The total duration of the trial was approximately 28 weeks for each individual participant, including the Follow-up. The participants received cebranopadol for a maximum of approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed indicating that the participant understands the purpose of and procedures required for the trial and is willing to participate in the trial.
* Participants must be at least 18 years of age at the Enrollment Visit.
* Women of childbearing potential must have a negative pregnancy test at enrollment and must not be lactating at the Enrollment Visit.
* Participants must be willing to use medically acceptable and highly effective methods of birth control.
* Participants who have completed treatment in KF6005/07 and are still in need of around-the-clock pain analgesia with strong opioids.

Exclusion Criteria:

* The participant has a clinically significant disease or condition other than cancer which in the investigator's opinion may affect efficacy or safety assessments.
* Known to or suspected of not being able to comply with the protocol and the use of cebranopadol.
* Participants taking forbidden concomitant medications or not being able to follow the rules of use of concomitant treatment.
* History of torsade de pointes and/or presence of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, bradycardia).
* Concurrent participation in another trial (except participation in KF6005/07) or planning to be enrolled in another clinical trial (i.e., administration of experimental treatment in another clinical trial) during the course of this trial, or previous participation in this trial.
* Employees of the sponsor, investigator, or trial site or family members of the employees, sponsor, or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (22):
- AT004, Vienna, Austria
- BE001, Sint-Niklaas, Belgium
- Bulgaria (4):
  - BG001, Shumen
  - BG008, Sofia
  - BG003, Sofia
  - BG004, Sofia
- Denmark (2):
  - DK006, Aalborg
  - DK004, Herlev
- Germany (2):
  - DE008, Böhlen
  - DE010, Munich
- HU011, Nyíregyháza, Hungary
- Poland (4):
  - PL012, Będzin
  - PL014, Dąbrowa Górnicza
  - PL003, Gdansk
  - PL010, Gliwice
- RO002, Cluj-Napoca, Romania
- Serbia (3):
  - RS003, Belgrade
  - RS002, Kamenitz
  - RS005, Zrenjanin
- Slovakia (3):
  - SK004, Bratislava
  - SK001, Prešov
  - SK005, Pruské

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koch ED, Kapanadze S, Eerdekens MH, Kralidis G, Letal J, Sabatschus I, Ahmedzai SH. Cebranopadol, a Novel First-in-Class Analgesic Drug Candidate: First Experience With Cancer-Related Pain for up to 26 Weeks. J Pain Symptom Manage. 2019 Sep;58(3):390-399. doi: 10.1016/j.jpainsymman.2019.05.012. Epub 2019 May 30. PMID 31152783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on the 18 Dec 2013 (first dose taken on the 19 Dec 2013 received) and the last participant completed the trial on the 03 May 2016 (last dose taken on the 12 Apr 2016). All participants in this trial completed the maintenance period in the KF6005/07 (NCT01964378) trial.
Pre-assignment Details: Participants who completed treatment in KF6005/07 and who were still in need of around-the-clock pain analgesia with strong opioids directly entered the KF6005/09 trial from the KF6005/07 trial. Seventy-six participants (37 previously on cebranopadol and 39 subjects previously on morphine treatment) were enrolled in this trial.
Groups:
- Cebranopadol: Cebranopadol: Cebranopadol 200 µg to 1000 µg per day taken once a day in the morning.
Period: Overall Study
Arm/Group | Cebranopadol
Started | 76
Completing the Titration Phase | 67
Completing the Treatment | 39
Completed | 38
Not Completed | 38
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 5
Not completed — Cancer Progression | 2
Not completed — Withdrawn as forbidden meds required | 1
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1
Not completed — Inclusion/Exclusion criteria not met | 5
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Population: Participants who completed treatment in KF6005/07 started on a daily dose of 200 or 400 μg (depending on previous dose level) in KF6005/09. The treatment code from KF6005/07 was not unblinded at the time of cebranopadol treatment initiation in KF6005/09, and in this trial all participants were titrated to their optimal dose of cebranopadol.
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.81)
Age, Customized [Count of Participants; unit: Participants]
  Below 18 years | 0
  From 18 to less than 65 years | 43
  From 65 to less than 85 years | 33
  Above 85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76
Region of Enrollment [Number; unit: participants]
  Romania | 2
  Hungary | 2
  Austria | 3
  Belgium | 1
  Denmark | 2
  Poland | 17
  Slovakia | 21
  Bulgaria | 4
  Serbia | 4
  Germany | 20
DN4 Neuropathic Pain at start of KF6005/07 [Number; unit: participants] — DN4 (Douleur Neuropathique en 4 Questions) was used as a screening tool for neuropathic pain. The DN4 consists of a total of 10 questions and tests, including interview questions (DN4-interview) and physical tests. The DN4 test was considered "positive" if there was a score of 4 or more (the maximum score is 10) then the participant has a neuropathic pain component. If the DN4 is negative, i.e., a score 3 or less then the participant was considered not to have a neuropathic pain component.
  participants
    DN4 positive | 21
    DN4 negative | 55
Height [Mean (Standard Deviation); unit: meter] | 1.684 (0.0844)
Weight [Mean (Standard Deviation); unit: kilograms] | 72 (14.04)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.36 (4.5)
Weekly means of average daily pain [Mean (Standard Deviation); unit: units on a scale] — For this assessment, each participant was asked "Please rate your pain by selecting the one number that best describes your pain on average during the last 24 hours" on an 11-point Numerical Rating Scale, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The mean of the assessments of average pain intensity in the last 24 hours in the last 3 days prior to first intake of cebranopadol is reported.
  units on a scale | 2.96 (1.89)
Weekly means of worst daily pain [Mean (Standard Deviation); unit: units on a scale] — For this assessment, each participant was asked "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 24 hours" on an 11-point Numerical Rating Scale, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The mean of the assessments of worst pain intensity in the last 24 hours in the last 3 days prior to first intake of cebranopadol is reported.
  units on a scale | 3.95 (2.447)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAEs)
Description: The safety of cebranopadol was assessed by the number of participants with treatment emergent adverse events (TEAEs). A TEAE was any adverse event that occurred after the first administration of investigational medicinal product (IMP), i.e., cebranopadol in this study. In addition, pretreatment adverse events which worsened during the treatment period were also considered TEAEs.
Time Frame: Up to 28 weeks (26 weeks of cebranopadol treatment and 2 weeks follow up after the last dose)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Groups:
- Cebranopadol: Cebranopadol (GRT6005) 200 µg to 1000 µg per day taken once a day in the morning.
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Participants | 64

2. Secondary Outcome: Intensity of Treatment Emergent Adverse Events
Description: A Treatment Emergent Adverse Event (TEAE) was defined as any Adverse Event (AE) that occurred on or after the first intake of cebranopadol or a pretreatment AE which worsened during the treatment period. TEAEs were classified by the investigator as falling into 1 of 3 categories:
  Mild: Signs and symptoms that can be easily tolerated. Symptoms can be ignored and disappear when the participant is distracted.
  Moderate: Symptoms cause discomfort but are tolerable; they cannot be ignored and affect concentration.
  Severe: Symptoms which affect usual daily activity.
  For TEAE where the intensity changed over time, the maximum intensity observed during the whole duration of the adverse event was documented.
Time Frame: Up to 28 weeks (26 weeks of cebranopadol treatment and 2 weeks follow-up after the last dose)
Population: Safety Set; event-based analysis
Measure: Number; unit: Number of TEAEs
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 661
Number of TEAEs
  Mild intensity | 242
  Moderate intensity | 300
  Severe intensity | 119

3. Secondary Outcome: Changes From Baseline in the Average Pain Intensity in the Last Week During the Treatment Period
Description: Participants were asked "Please rate your pain by selecting the one number that best describes your pain on average during the last week." and scored their average pain intensity during the last week of the treatment period on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The absolute change from baseline for the average pain intensity during the last week was determined for all participants that scored their pain intensities. A mean value for all participants was calculated.
Time Frame: Baseline Visit (Day 1) to End of Treatment Visit (up to 26 weeks).
Population: Safety Set - participants with data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 59
units on a scale | 0.8 (2.14)

4. Other Pre Specified Outcome: Outcome of Treatment Emergent Adverse Events (TEAE)
Description: The outcome of a TEAE was classified into 1 of the following 6 categories by the investigator, i.e.
  * Recovered/Resolved.
  * Recovered/Resolved with sequelae.
  * Fatal
  * Recovering/Resolving.
  * Not recovered/Not resolved.
  * Unknown (e.g., because the participant is lost to follow up).
Time Frame: Baseline (Day 2) to End of trial (i.e., up to Week 28)
Population: Safety Set; event-based analysis
Measure: Number; unit: Number of TEAEs
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 661
Number of TEAEs
  Recovered/resolved | 349
  Recovered/resolved with sequelae | 11
  Not recovered/not resolved | 260
  Recovering/resolving | 14
  Fatal | 11
  Unknown | 16

5. Other Pre Specified Outcome: Time to Onset of Treatment Emergent Adverse Events (TEAEs)
Description: The median time, in days, from the start of the open-label cebranopadol treatment to the start day of the treatment emergent adverse event (TEAE).
Time Frame: Baseline (Day 2) to End of trial (up to Week 28)
Population: Safety Set; event-based analysis for 661 TEAEs.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 661
days | 53.0 [19 to 106]

6. Other Pre Specified Outcome: Duration of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence attributed to cebranopadol. Duration of Adverse Event was calculated as stop date minus start date plus 1 for non-missing and partial dates.
Time Frame: Baseline (Day 2) to End of trial (up to Week 28)
Population: Safety Set; data available for 373 TEAEs (duration data for 288 of 661 TEAEs were not available)
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 373
days | 9.0 [3 to 27]

7. Other Pre Specified Outcome: Causal Relationship of Treatment Emergent Adverse Events (TEAEs)
Description: The causality of TEAEs was assessed by the investigator as falling into 1 of the following 7 categories: Conditional/Unclassified, Unassessable/Unclassifiable, Not related, Unlikely, Possible, Probable/likely, or Certain. The numbers of TEAEs per category are presented.
Time Frame: Baseline (Day 2) to End of trial (up to Week 28)
Population: Safety Set; event-based analysis on 661 TEAEs
Measure: Number; unit: Number of TEAEs
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 661
Number of TEAEs
  Certainly Related | 0
  Possibly Related | 42
  Probably/Likely Related | 7
  Unlikely Related | 37
  Not Related | 574
  Unassessable/Unclassifiable | 1
  Conditional/Unclassifiable | 0

8. Other Pre Specified Outcome: Countermeasures Taken for Treatment Emergent Adverse Events (TEAEs)
Description: The countermeasure of a Treatment Emergent Adverse Event (TEAE) was classified by the investigator as being a study medication-related countermeasure and based on non-study medication countermeasures.
  Non-study medication related countermeasures were categorized as being one of the following: No countermeasure given; A newly started medication or change in dose or route of application of a concomitant medication due to the AE; Other countermeasures, e.g., physical therapy, surgery.
  Study medication-related countermeasures were categorized as being one of the following: Dose not changed; Dose reduced; Drug interrupted; Trial discontinuation.
  Absolute numbers are per category reported.
Time Frame: Baseline (Day 2) to End of trial (up to Week 28)
Population: Safety Set; event-based analysis.
Measure: Number; unit: Number of TEAEs
Units Other Than Participants: Number of TEAEs
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Number analyzed (Number of TEAEs) | 661
Number of TEAEs
  No countermeasure | 361
  Newly started medication | 281
  Other | 19
  Cebranopadol dose not changed as countermeasure | 595
  Cebranopadol dose reduced | 5
  Cebranopadol treatment interrupted | 14
  Cebranopadol withdrawn | 23
  Cebranopadol to dosing missing | 24

9. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Related to Cebranopadol
Description: Only participants with TEAEs which were assessed by the investigator as falling into one of the 3 categories of causality (Possible, Probable/likely, or Certain) were summarized. The initial breakdown planned based on intensity, outcome, time to onset, duration, and countermeasures was not performed and is therefore not reported.
Time Frame: Baseline (Day 2) to End of trial (up to Week 28)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Participants
  Participants with related TEAEs | 20
  Participants with related serious TEAEs | 1
  Participants without related TEAEs | 55

10. Other Pre Specified Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) Scores
Description: The C-SSRS was administered by a clinician who had been certified to administer the C-SSRS at each visit. Suicidal ideation is classified on a 5-item scale (where 1 = Wish to be dead, 2 = Non-specific active suicidal thoughts, 3 = Active Suicidal Ideation with any methods (not plan) without intent to act, 4 = Active Suicidal Ideation with some intent to act, without specific plan, 5 = Active suicidal ideation with a specific plan and intent). The number of participants with suicidal ideation at baseline is presented below for categories with at least 1 participant.
Time Frame: Baseline (Day 1) to End of trial (up to Week 28)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Participants
  No suicidal ideation or behaviour | 74
  Wish to be dead | 1
  Non-specific active suicidal thoughts | 1

11. Other Pre Specified Outcome: Mean Scores of Chronic Pain Sleep Inventory (CPSI) and Changes From Baseline
Description: The CPSI was completed by the participants. It measures 5 items, all on a 100-mm visual analog scale:
  Participant's assessment of Sleep Problem Index subscores and need for sleep medication (the lower the score the better): (1) Trouble falling asleep (0 = never; 100 = always); (2) Needing sleep medication to help fall asleep (0 = never, 100 = always); (3) Awakened by pain during the night (0 = never, 100 = always); and (4) Awakened by pain in the morning (0 = never, 100 = always). The Sleep Problem Index is the sum of items (1), (3), and (4) with a maximum score of 100 indicating maximum sleep problems.
  Participant's assessment of the Overall Quality of Sleep (the higher the score the better): (5) Overall quality of sleep (0 = very poor, 100 = excellent).
Time Frame: Baseline (Day 1); End of Treatment (up to Week 26)
Population: Safety Set; participants with data available at respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline - Trouble falling asleep | 10.0 (18.00)
  End of Treatment - Trouble falling asleep: number analyzed (Participants) | 58
  End of Treatment - Trouble falling asleep | 11.7 (22.91)
  Baseline - Need for sleep medication | 9.2 (24.93)
  End of Treatment - Need for sleep medication: number analyzed (Participants) | 58
  End of Treatment - Need for sleep medication | 10.7 (28.53)
  Baseline - Woken up by pain during night | 12.5 (21.02)
  End of Treatment - Woken up by pain during night: number analyzed (Participants) | 58
  End of Treatment - Woken up by pain during night | 15.3 (26.36)
  Baseline - Woken by pain in the morning | 12.6 (20.71)
  End of Treatment - Woken by pain in the morning: number analyzed (Participants) | 58
  End of Treatment - Woken by pain in the morning | 17.5 (28.21)
  Baseline - Overall quality of sleep | 74.0 (27.91)
  End of Treatment - Overall quality of sleep: number analyzed (Participants) | 58
  End of Treatment - Overall quality of sleep | 71.3 (30.97)
  Baseline - Sleep Problem Index | 35.0 (54.03)
  End of Treatment - Sleep Problem Index: number analyzed (Participants) | 58
  End of Treatment - Sleep Problem Index | 44.5 (71.10)

12. Other Pre Specified Outcome: Weekly Means of Daily Average Pain Intensity During the First Month of Treatment
Description: Participants were asked: "Please rate your pain by selecting the one number that best describes your pain on average during the last 24 hours." every day in the morning during the first month of treatment (comprising Titration Weeks 1 and 2 and Maintenance Weeks 1 and 2). They scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The weekly mean value of the 24-hour average pain intensity was calculated as a mean score of these daily entries of average pain intensity for each week.
Time Frame: Baseline (Day 1); Titration Weeks 1 and 2; Maintenance Weeks 1 and 2
Population: Safety Set; data for participants who completed respective visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline | 2.96 (1.890)
  Titration Week 1 | 3.18 (1.795)
  Titration Week 2: number analyzed (Participants) | 68
  Titration Week 2 | 2.90 (1.838)
  Maintenance Week 1: number analyzed (Participants) | 66
  Maintenance Week 1 | 2.73 (1.848)
  Maintenance Week 2: number analyzed (Participants) | 66
  Maintenance Week 2 | 2.69 (1.843)

13. Other Pre Specified Outcome: Worst Pain Intensity in the Last Week of Treatment (Week 26)
Description: Participants were asked: "Please rate your pain by selecting the one number that best describes your pain at its worst during the last week." at some of the visits during the treatment period. They scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The mean scores of the worst pain intensity were calculated for all participants. Results for baseline and Week 26 are presented.
Time Frame: Baseline (Day 1); End of Treatment (Week 26)
Population: Safety Set; 59 participants completed End of Treatment Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline | 4.3 (2.52)
  End of Treatment (Week 26): number analyzed (Participants) | 59
  End of Treatment (Week 26) | 5.1 (2.89)

14. Other Pre Specified Outcome: Weekly Average Number of Breakthrough Pain Episodes
Description: The number of episodes of breakthrough pain during the past week was planned to be collected. However, for some participants, the intensity of breakthrough pain for the past week has been collected instead of the incidence of breakthrough pain events. Since the values of the intensity of breakthrough pain were much higher (maximum of up to 99) than the frequency of pain events, the mean is skewed and cannot be interpreted. The median for the weekly average number of breakthrough pain episodes is less influenced by these values and is reported below.
Time Frame: Baseline (Day 1); End of Treatment (Week 26)
Population: Safety Set; 61 participants completed End of Treatment Visit
Measure: Median (Full Range); unit: Weekly average number of episodes
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
Weekly average number of episodes
  Baseline | 1.00 [0.0 to 66.0]
  End of Treatment (Week 26): number analyzed (Participants) | 61
  End of Treatment (Week 26) | 1.00 [0.0 to 99.0]

15. Other Pre Specified Outcome: Mean Scores of Neuropathic Pain Symptom Inventory (NPSI)
Description: Participants with neuropathic pain (determined by the completion of the DN4 [Douleur Neuropathique] questionnaire at enrollment) rated their symptoms of neuropathic pain using the NPSI. Ten out of 12 questions (Q1-3, 5, 6, 8-12) are answered on an 11-point numerical scale (NRS) ranging from 0 (no symptom present) to 10 (worst imaginable).
  The NPSI Total Score was calculated as the sum of the 10 single items scored on the 11-point NRS divided by 100. The mean score is reported on a scale of 0 (no neuropathic pain components present) to 1 (all neuropathic pain components have the maximum imaginable intensity).
Time Frame: Baseline (Day 1); Weeks 2, 6, 14, 18; End of Treatment (up to Week 26)
Population: Safety Set (21 participants with neuropathic pain of 76 participants enrolled)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 21
units on a scale
  Baseline | 0.243 (0.1677)
  Week 2: number analyzed (Participants) | 20
  Week 2 | 0.200 (0.2006)
  Week 6: number analyzed (Participants) | 16
  Week 6 | 0.146 (0.1397)
  Week 14: number analyzed (Participants) | 10
  Week 14 | 0.150 (0.1564)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 0.117 (0.1529)
  Final Visit (Week 26): number analyzed (Participants) | 11
  Final Visit (Week 26) | 0.236 (0.2183)

16. Other Pre Specified Outcome: EuroQol-5 Dimension (EQ-5D) Health Status Index Outcome
Description: Participants answered 5 questions on the 5 dimensions of the EuroQol-5 Dimension Health Questionnaire: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each question has 3 possible answers reflecting 3 levels of impact on the quality of life. Each dimension was assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the 5 EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D Health Status Index score between 0 to 1 (with 1 indicating "full health" and 0 representing "dead"). The higher the values (the closer the value is to 1), the better the health status.
Time Frame: Baseline (Day 1); End of Treatment (up to Week 26)
Population: Safety Set; participants with data available at respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline: number analyzed (Participants) | 75
  Baseline | 0.687 (0.2111)
  Final Visit (Week 26): number analyzed (Participants) | 58
  Final Visit (Week 26) | 0.606 (0.3214)

17. Other Pre Specified Outcome: EuroQol-5 Dimension (EQ-5D) Health Questionnaire - Visual Analog Scale (VAS)
Description: The EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant-rated scale where a single value is ticked for "Your own health state today" on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline (Day 1); End of Treatment (up to Week 26)
Population: Safety Set; participants with data available at respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline: number analyzed (Participants) | 74
  Baseline | 61.9 (20.62)
  Final Visit (Week 26): number analyzed (Participants) | 58
  Final Visit (Week 26) | 56.6 (21.94)

18. Other Pre Specified Outcome: Patient Global Impression of Change (PGIC)
Description: In the PGIC, participants indicates the perceived change over the treatment period compared to their condition prior to the start of treatment. Participants are requested to choose 1 of 7 categories. Scores range from "very much improved" to "very much worse". The frequency of responses per category are provided.
Time Frame: Baseline (Day 1); End of Treatment (up to Week 26)
Population: Safety Set; 62 participants completed the End of Treatment Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol
Number analyzed (Participants) | 62
Participants
  Very much improved | 5
  Much improved | 17
  Minimally improved | 15
  No change | 9
  Minimally worse | 8
  Much worse | 3
  Very much worse | 1
  Missing | 4

19. Other Pre Specified Outcome: Clinical Global Impression of Change (CGIC)
Description: For the CGIC assessment, the clinician indicates the perceived change in the patient's condition over the treatment period as compared to the patient's condition prior to the start of treatment. The clinician is requested to choose 1 of 7 categories. Categories range from "very much improved" to "very much worse".
Time Frame: Baseline (Day 1); End of Treatment Visit (up to Week 26)
Population: Safety Set; 62 participants completed the End of Treatment Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cebranopadol
Number analyzed (Participants) | 62
Participants
  Very much improved | 9
  Much improved | 25
  Minimally improved | 10
  No change | 5
  Minimally worse | 4
  Much worse | 3
  Very much worse | 3
  Missing | 3

20. Other Pre Specified Outcome: Use of On-demand Opioid Analgesic Medication
Description: Participants reported the opioid type and amount of an opioid in mg/day used to relieve their breakthrough pain over the time period in the study. The average number of units of on-demand opioid medication administered during the previous day (reported on Day 3) and during the last 3 days (reported at all other visits) were documented. The number of units of on-demand opioid medication administered during the Treatment Period is summarized descriptively over the treatment period.
Time Frame: From Day 3 to End of Treatment (up to Week 26) (13 time points)
Population: Safety Set; participants with data available at the respective visit.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units
  Day 3 | 1.08 (1.772)
  Week 1: number analyzed (Participants) | 68
  Week 1 | 1.45 (2.396)
  Day 11: number analyzed (Participants) | 68
  Day 11 | 1.29 (2.280)
  Week 2: number analyzed (Participants) | 68
  Week 2 | 0.96 (1.817)
  Day 17: number analyzed (Participants) | 67
  Day 17 | 0.64 (1.218)
  Week 3: number analyzed (Participants) | 67
  Week 3 | 0.78 (2.126)
  Week 4: number analyzed (Participants) | 64
  Week 4 | 0.72 (1.380)
  Week 6: number analyzed (Participants) | 63
  Week 6 | 0.59 (1.252)
  Week 10: number analyzed (Participants) | 52
  Week 10 | 0.51 (1.044)
  Week 14: number analyzed (Participants) | 49
  Week 14 | 0.47 (1.174)
  Week 18: number analyzed (Participants) | 45
  Week 18 | 0.55 (1.250)
  Week 22: number analyzed (Participants) | 43
  Week 22 | 0.77 (1.641)
  End of Treatment (up to Week 26): number analyzed (Participants) | 62
  End of Treatment (up to Week 26) | 1.06 (2.397)

21. Other Pre Specified Outcome: Mean Equipotency Ratio of Morphine Sulfate Prolonged Release Compared to Cebranopadol.
Description: For those participants, who received morphine prolonged release in the CORAL trial (KF6005/07, NCT01964378) and were, thus, switched from morphine prolonged release to cebranopadol in the CORAL XT trial, the equianalgesic doses of morphine prolonged release and cebranopadol was identified.
Time Frame: Baseline (Day 1); End of first month of treatment
Population: Safety Set; the Conversion Ratio of Morphine Prolonged Release to Cebranopadol was available for 32 of 76 participants.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cebranopadol
Number analyzed (Participants) | 32
Ratio | 156.8 (58.2)

22. Other Pre Specified Outcome: Mean Eastern Cooperative Oncology Group Performance Status (ECOG) Scores
Description: The investigator scores the ECOG performance status for a participant on a 6-point categorical scale as follows:
  * 0 indicates that a participant is "fully active, able to carry on all pre-disease performance without restriction."
  * 1 indicates that a participant is "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work."
  * 2 indicates that a participant is "ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours."
  * 3 indicates that a participant is "capable of only limited selfcare, confined to bed or chair more than 50% of waking hours."
  * 4 indicates that a participant is "completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair."
  * 5 indicates that a participant is "dead". Mean ECOG performance status scores are calculated for the number of participants with data available.
Time Frame: From Baseline (Day 1) through to End of treatment (up to Week 26) (9 time points)
Population: Safety Set; number of participants with data available at the respective visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cebranopadol
Number analyzed (Participants) | 76
units on a scale
  Baseline | 1.1 (0.75)
  Week 2: number analyzed (Participants) | 67
  Week 2 | 1.1 (0.76)
  Week 4: number analyzed (Participants) | 64
  Week 4 | 1.1 (0.78)
  Week 6: number analyzed (Participants) | 63
  Week 6 | 1.2 (0.74)
  Week 10: number analyzed (Participants) | 52
  Week 10 | 1.1 (0.77)
  Week 14: number analyzed (Participants) | 49
  Week 14 | 1.1 (0.73)
  Week 18: number analyzed (Participants) | 45
  Week 18 | 1.2 (0.91)
  Week 22: number analyzed (Participants) | 42
  Week 22 | 1.4 (0.82)
  Final Visit (up to Week 26): number analyzed (Participants) | 63
  Final Visit (up to Week 26) | 1.6 (1.10)

ADVERSE EVENTS:
Time Frame: All AEs were documented from the time of enrollment (i.e., the time the informed consent form was signed) up to the time of the last protocol scheduled contact occurred, i.e., date of last visit/contact (a telephone call in the case of discontinuation). Treatment emergent adverse events (TEAEs) were reported for up to 28 weeks (26 weeks of cebranopadol treatment and 2 weeks follow-up after the last dose).
Description: Tables below present TEAEs reported in participants who took at least 1 dose of cebranopadol (Safety Set).
  Ten participants died during the trial; 5 further deaths occurred after the participants were discontinued from the trial and were reported spontaneously by the investigators.
Groups:
- Cebranopadol: Cebranopadol: Cebranopadol 200 µg to 1000 µg per day taken once a day in the morning.
  Subjects who completed the treatment in KF6005/07 and were willing to participate in this trial went into a Titration Phase (approximately 2 weeks). During the Titration Phase, the subjects were titrated to their individual optimal daily dose of cebranopadol, defined as a balance between self-reported analgesia and side effects.
Arm/Group | Cebranopadol
All-Cause Mortality (participants affected / at risk) | 10/76
Serious Adverse Events (participants affected / at risk) | 32/76
Other Adverse Events (participants affected / at risk) | 63/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cebranopadol (N=76)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (26)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asthenia (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Facial bone fracture (Injury, poisoning and procedural complications) | 1 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Epilespsy (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cebranopadol (N=76)
Gamma-glutamyltransferase increased (Investigations) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytosis (Blood and lymphatic system disorders) | 7 (10)
Headache (Nervous system disorders) | 8 (8)
Somnolence (Nervous system disorders) | 8 (9)
Dizziness (Nervous system disorders) | 5 (6)
Asthenia (General disorders) | 19 (21)
Fatigue (General disorders) | 9 (10)
Feeling drunk (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 9 (9)
Pyrexia (General disorders) | 9 (10)
Depressed mood (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (7)
Nervousness (Psychiatric disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 17 (21)
Bacteriuria (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (7)
Nausea (Gastrointestinal disorders) | 15 (18)
Vomiting (Gastrointestinal disorders) | 8 (11)

LIMITATIONS AND CAVEATS:
A limitation is the open-label design of the study. An extrapolation to a population not suffering from cancer-related pain is limited due to the nature of the underlying disorder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.